CLINICAL TRIAL: NCT00739167
Title: A Quality of Life Study for Patients With Primary or Metastatic Liver Cancer Who Are Treated With Radioembolization (Y90 Microspheres) or Transcatheter Arterial Embolization (TACE)
Brief Title: Quality of Life in Patients Undergoing Embolization Using Yttrium Y 90 Glass Microspheres for Primary or Metastatic Liver Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NU 07Q1; P30CA060553 (NIH); NU-07Q1; NU-IRB-STU00002799
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; liver metastases; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Y90 Group: Patients receiving treatment with radioembolization.
- TACE Group: Patients receiving treatment with transcatheter arterial embolization
- RFA Group: Patients receiving treatment with radiofrequency ablation.

SUMMARY:
RATIONALE: Learning about quality of life in patients with cancer undergoing embolization may help doctors learn about the side effects of treatment and plan the best treatment.

PURPOSE: This clinical trial is studying quality of life in patients undergoing embolization using yttrium Y 90 glass microspheres for primary or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the quality of life (QOL) as defined by the presence or absence of physical, social, emotional, and functional distress in patients with primary or metastatic liver cancer undergoing treatment with radioembolization or transcatheter arterial embolization.
* Compare the time course of QOL measures between treatment groups in patients treated with these regimens.
* Compare the time course of QOL measures between patient subgroups defined by pre-treatment quality of life or tumor burden.

OUTLINE: Patients complete FACT-Hep version 4 surveys on quality of life prior to initiation of embolization, and at 2 weeks and 1 month after completion of embolization.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary hepatocellular cancer or metastatic liver cancer
* Planning radioembolization or transcatheter arterial embolization using yttrium Y 90 glass microspheres
* No encephalopathy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Bilirubin ≤ 3 mg/dL
* Able to comply with study procedures

PRIOR CONCURRENT THERAPY:

* No prior treatment with radioembolization or transcatheter arterial embolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of hepatocellular carcinoma being treated with either TACE, RFA, or Y90.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Quality of life of all patients over the course of treatment | Before treatment, 2 weeks post, and 1 month post
Quality of life differences between treatment groups | Before treatment, 2 weeks post, and 1 month post

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Gilbertsen, RN, BS, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Salem R, Gilbertsen M, Butt Z, Memon K, Vouche M, Hickey R, Baker T, Abecassis MM, Atassi R, Riaz A, Cella D, Burns JL, Ganger D, Benson AB 3rd, Mulcahy MF, Kulik L, Lewandowski R. Increased quality of life among hepatocellular carcinoma patients treated with radioembolization, compared with chemoembolization. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1358-1365.e1. doi: 10.1016/j.cgh.2013.04.028. Epub 2013 May 2. PMID 23644386